CLINICAL TRIAL: NCT01149759
Title: Evaluate Reversal of Pathological Epidermal Phenotype in Severe Atopic Dermatitis With Suppression of Immune Activation During Cyclosporine Therapy
Brief Title: Reversal of Epidermal Phenotype in Severe Atopic Dermatitis With Cyclosporine Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Principal Investigator, Mary Sullivan-Whalen, Research Nurse Practictioner, Rockefeller University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JKR-0663
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Atopic Dermatitis; Eczema
Keywords: Atopic Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cyclosporine A (Experimental): 5 mg/kg for first 4 weeks, followed by tapering to 1 mg/kg for 12 weeks until discontinuation at 16 weeks.
  Interventions: Drug: Cyclosporine A

INTERVENTIONS:
Drug: Cyclosporine A — 5 mg/kg for first 4 weeks, followed by tapering to 1 mg/kg for 12 weeks until discontinuation at 16 weeks
  Other Names: Neoral

SUMMARY:
Atopic Dermatitis (AD) or eczema is a chronic relapsing inflammatory disease that affects 1-3% of the adults and up to 25% of the children in the United States. Patients with severe AD will be studied during a 24-week study with systemic cyclosporine (Neoral, capsule form) to evaluate the immune suppression and pathological correlation of cyclosporine A in these patients in order to determine the extent to which immune activation drives the pathological epidermal phenotype.

DETAILED DESCRIPTION:
Patients will be first screened to be sure they are healthy (aside from atopic dermatitis) with a physical exam, and lab tests. These lab tests consist of CBC, biochemical profile, hepatitis B and C profile, urine analysis, HIV, PPD, and urine pregnancy test (if applicable). Patients will return in 2 to 3 days for PPD reading. A repeat serum creatinine will be drawn at this time so as to have 2 baseline values. Patient will begin taking cyclosporine at 5 mg/kg of body weight in 2 divided daily doses for 12 weeks, and after this period the dose will be reduced by 1mg/kg per week (the tapering down will start at 12 weeks of treatment), so that cessation of treatment will occur after 16 weeks from the start of treatment. Patients will then be followed in clinic for an additional 8 weeks for a potential relapse, and if a relapse will occur topical treatment with corticosteroids, immune-modulators or phototherapy may be instituted. Patients will be seen in the outpatient clinic at baseline, wks 1,2, 4, 6, 8, 10, and 12 and every 2weeks until completion of a 24-week study. Biopsies (of lesional and non-lesional skin) will be done to assess histological response at baseline, week 2, week 6 (optional), week 12 and at relapse (optional). Bloods for safety analysis and pregnancy test (if applicable) will be done at each visit, and vital signs will be measured at that time. Serum IgE, eosinophils, and serum cytokines will be done at baseline, and every 2 weeks until week 16, and at week 24. At each visit patients will be assessed for adverse events. Clinical assessment, and ultrasound, will be done at each visit. The most widely accepted clinical assessment tool is known as SCORAD (SCORing for Atopic Dermatitis). This tool combines clinical features of AD such as erythema, dryness, lichenification, percent body surface area, as well as quality of life issues such as pruritus and loss of sleep due to disease. Another assessment tool we will be using is the static IGA (investigator global assessment). The IGA represents an overall evaluation of dermatitis performed by the investigator at every visit. IGA scores utilize a 6-point scale, ranging from 0 (clear) to 5 (very severe disease). IGA scores measure disease severity based on morphology, without referring back to the baseline state. Ultrasound study provides an alternate, non-invasive method of assessing disease activity in the skin. Clinical photos will be done at weeks 0, 6, 12, 16, and 24.In this study, we would like to determine whether AD, like psoriasis, is an immune-driven disease of epidermal hyperplasia and differentiation. To establish the immune contribution to AD, we will treat patients with standard doses of CsA and measure the extent of immune suppression in skin lesions by quantitative measures of pathological leukocytes and expression of inflammatory gene products. At the end of 12 weeks of treatment we will determine whether pathological epidermal hyperplasia is reversed by quantitative and qualitative measures of epidermal hyperplasia and aberrant epidermal differentiation. In addition, we will correlate the extent to which the epidermal phenotype is modulated with the extent to which skin inflammation is suppressed, as the effect of suppression of specific inflammatory molecules on resulting keratinocyte responses is not known. The alternative hypothesis in AD is that it is not an immune-mediated disease, but instead a disease of primary epidermal differentiation due to germline alterations (gene deletions) in filaggrin and other genes that cooperate to differentiate a normal epidermal barrier at the level of stratum corneum. The alternative hypothesis is considered to be the most likely patho-mechanism in AD by a number of current researchers. The alternative hypothesis would be supported by this study if pathologic epidermal hyperplasia persists in the skin regions with significant suppression of the immune/inflammatory pathways induced by CsA treatment.

ELIGIBILITY:
Inclusion Criteria:

* Severe AD (defined as having a mean SCORAD score> 40,, with significant disease activity, pruritus, and sleep disturbances (13), suitable for treatment with Cyclosporine, and have failed or unsuitable for other treatment modalities, including topical and or systemic steroids or phototherapy. Patients must also have an IGA score of 3 or greater,
* Males and females age 18 and above (if females are of child-bearing potential they must agree to use acceptable contraception during the study).
* No systemic treatment contraception must commence 2 weeks prior to initiating the drug.
* No systemic treatment for 4 weeks, no topical treatment or phototherapy for 2 weeks

Exclusion Criteria:

* Previously treated with cyclosporine and had unacceptable toxicity
* Past or current history of malignancy (except for treated isolated skin cancers)
* Renal, hepatic, and hematologic laboratory values greater than CTC grade 1 toxicity, such as but not limited to creatinine >1.5 ULN, SGOT>2.5 ULN. Values greater then grade 1 would most likely represent clinically significant renal, hepatic or hematologic disease
* Stage I hypertension is defined as >140/90. Patients with this blood pressure or higher on two separate occasions, whether on medications or not, will be excluded (JNC guidelines www.nhlbi.nih.gov/guidelines/hypertension )
* Significant lipid panel abnormality (any grade 1 toxicity on CTC scale)
* Lactating females
* Other medical condition that would increase the risk of cyclosporine toxicity
* Positive PPD
* Primary or secondary immune deficiency (including known HIV status)
* Possible or known pregnancy
* Serious infection (such as active hepatitis)
* Drug or alcohol abuse
* Inability or lack of willingness to co-operate with regular monitoring
* Severe photodamage/precancerous skin lesions due to previous sunlight exposure, or photo/photochemotherapy
* Concurrent use of PUVA or UVB, other radiation therapy,
* Concurrent use of other immunosuppressive agents such as MTX, Immuran, Cyclophosphamide, Cellcept, etc.(because of the possibility of excessive immunosuppression and the subsequent risk of malignancies)
* Active infections, infections or history of serious infection requiring hospitalization, antibiotics, antivirals,or antifungals within 30 days of baseline
* History of other inflammatory skin conditions (such as psoriasis, pemphigus, etc.
* Patients with background skin conditions that might be directly related to atopic dermatitis (such as post inflammatory hyperpigmentation) will not be excluded as well as common background non-inflammatory skin conditions such as seborrheic keratosis, benign pigmented lesions, acne, etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Krueger, MD, PhD, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cyclosporine A
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cyclosporine A
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: SCORAD Change Score
Description: SCORAD ("SCORing Atopic Dermatitis") is a clinical tool for assessing the severity (i.e., extent, intensity) of atopic dermatitis (AD) as objectively as possible with scores ranging from 0-100. The higher the score indicates more severe AD. For this outcome the SCORAD change score is computed as an absolute number which is comparing improvement in the SCORAD score of participants at week 12 compared to their SCORAD score at baseline.
Time Frame: 12 weeks
Population: 9 were included in this analysis from Rockefeller University
Measure: Mean (Standard Deviation); unit: Change Score
Arm/Group | Cyclosporine A
Number analyzed (Participants) | 9
Change Score | 33.34 (19.87)

2. Secondary Outcome: Change in Epidermal Thickness
Description: Change in lesional skin epidermal thickness at week 12 compared to baseline
Time Frame: 12 weeks
Population: 9 participants were included in this analysis from Rockefeller University, this is a change in the skin thickness at week 12 compared to baseline
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Cyclosporine A
Number analyzed (Participants) | 9
micrometer | 79.70 (21.18)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Cyclosporine A
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No